CLINICAL TRIAL: NCT07381439
Title: A Prospective, Randomized Controlled Trial Comparing Conventional Linear Versus Novel Spiral Iodine-125 Seed Strand Implantation Combined With Metallic Stent for Malignant Obstructive Jaundice
Brief Title: Comparison of Two Seed Strand Implantation Techniques for Biliary Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Peng, Zhaohong, Associate Chief Physician, The First Affiliated Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LLSC20221301
Record Dates: First submitted 2026-01-14; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Malignant Obstructive Jaundice
Keywords: Malignant obstructive jaundice; 125I seeds strand; Complications

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group, randomized controlled trial comparing a novel spiral seed strand implantation technique with the conventional linear technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional linear implantation (Experimental): In this group, participants received percutaneous transhepatic biliary stenting combined with a straight-configured ^125^I seed strand. The strand was fabricated by loading the prescribed number of ^125^I seeds into a 4F catheter, the ends of which were subsequently heat-sealed. During the procedure, after the deployment of a self-expanding metallic stent across the malignant stricture, the straight seed strand was implanted and fixed in the space between the outer wall of the stent and the bile duct wall to deliver localized brachytherapy.
  Interventions: Radiation: Percutaneous transhepatic biliary stenting with conventional linear ^125^I seeds strand
- Novel spiral implantation (Experimental): In this group, participants received percutaneous transhepatic biliary stenting combined with a spiral-configured ^125^I seed strand. The strand was fabricated by first preparing a linear catheter strand and then shaping it into a spiral configuration using boiling water. A slightly higher number of seeds were used to compensate for foreshortening. During the procedure, after stent deployment, the spiral seed strand was implanted and secured within the inner lumen of the metallic stent. This method was designed to reduce tract-related injury by utilizing a single, smaller working sheath and minimizing manipulation of the bile duct wall.
  Interventions: Radiation: Percutaneous transhepatic biliary stenting with novel spiral ^125^I seeds strand

INTERVENTIONS:
Radiation: Percutaneous transhepatic biliary stenting with conventional linear ^125^I seeds strand — This is a combined interventional radiology procedure for malignant obstructive jaundice. Under local anesthesia and fluoroscopic guidance, a self-expanding metallic biliary stent is percutaneously placed across the malignant stricture. Subsequently, a linear strand of Iodine-125 (^125^I) seeds, fabricated by sealing the prescribed number of seeds within a catheter, is implanted and fixed in the space between the outer wall of the stent and the bile duct wall. The ^125^I seeds provide continuous low-dose-rate brachytherapy to inhibit tumor ingrowth and prolong stent patency.
  Other Names: PTBSIS
  Arms: Conventional linear implantation
Radiation: Percutaneous transhepatic biliary stenting with novel spiral ^125^I seeds strand — This is a combined interventional radiology procedure for malignant obstructive jaundice. Under local anesthesia and fluoroscopic guidance, a self-expanding metallic biliary stent is percutaneously placed across the malignant stricture. Subsequently, a spiral-configured strand of Iodine-125 (^125^I) seeds, fabricated by shaping a linear catheter strand with boiling water (using a slightly higher seed count to compensate for foreshortening), is implanted and secured within the inner lumen of the stent. The ^125^I seeds provide continuous low-dose-rate brachytherapy to inhibit tumor ingrowth and prolong stent patency. This method is designed to reduce tract-related injury by minimizing bile duct wall manipulation.
  Other Names: PTBSIS (novel)
  Arms: Novel spiral implantation

SUMMARY:
This study aimed to compare the safety and effectiveness of two different methods for fabricating and implanting Iodine-125 (^125^I) radioactive seed strands combined with a metal stent for treating malignant obstructive jaundice. The conventional method uses a straight seed strand placed between the stent and the bile duct wall. A novel technique was developed that uses a spiral-shaped seed strand placed inside the stent lumen.

Between January 2018 and February 2024, 105 patients were randomly assigned to two groups. Group A (59 patients) received the conventional straight strand, while Group B (46 patients) received the novel spiral strand. The study compared therapeutic efficacy, the incidence of intraoperative and postoperative complications, stent patency duration, and patient survival.

Both methods successfully improved liver function. However, the novel spiral technique (Group B) caused significantly fewer complications, such as bile leakage and peritonitis, compared to the conventional method (Group A). Importantly, patients in Group B also had longer stent patency (305 days vs. 277 days) and longer overall survival (345 days vs. 300 days).

In conclusion, the novel spiral seed strand implantation technique is a safer and more effective treatment option for malignant obstructive jaundice.

DETAILED DESCRIPTION:
Malignant obstructive jaundice often requires palliative drainage with self-expanding metallic stents. Combining stents with brachytherapy using Iodine-125 (^125^I) seed strands has been shown to prolong stent patency and patient survival compared to stenting alone. The conventional technique implants a linear seed strand between the stent and the bile duct wall, which is associated with risks of hemobilia, biliary fistula, and peritonitis due to the need for a larger puncture tract. This prospective, randomized controlled trial aimed to evaluate a novel, refined method involving a spiral-configured ^125^I seed strand implanted within the stent lumen, hypothesizing that it would reduce procedure-related complications while maintaining or improving therapeutic efficacy.

Study Design and Methods:

This was a single-center, prospective, randomized controlled trial. From January 2018 to February 2024, 105 patients with inoperable malignant obstructive jaundice were enrolled and randomly allocated into two groups.

Group A (Conventional, n=59): Received a straight ^125^I seed strand implanted between the metallic stent and the bile duct wall.

Group B (Novel, n=46): Received a spiral ^125^I seed strand implanted within the lumen of the metallic stent.

All patients first underwent percutaneous transhepatic biliary drainage (PTBD) for decompression, followed by the combined stent and seed strand (PTBSIS) procedure 3-7 days later.

Primary and Secondary Outcomes:

The primary endpoints were procedure-related complications (intraoperative and postoperative) and stent patency time. Secondary endpoints included technical success rate, improvement in liver function tests at one month, and overall patient survival. Complications assessed included nausea/vomiting, abdominal pain, hemobilia, vagal reflex, fever, biliary fistula, and biliary peritonitis.

Statistical Analysis:

Continuous data are presented as mean ± standard deviation or median (interquartile range). Categorical variables were compared using the Chi-square or Fisher's exact test. Stent patency and overall survival were analyzed using the Kaplan-Meier method with the log-rank test. A two-sided P-value < 0.05 was considered statistically significant. Analyses were performed using SPSS version 22.0.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with a definitive diagnosis of Malignant Obstructive Jaundice (MOJ) confirmed by imaging (enhanced CT/MRCP), laboratory tests, and/or pathology.

  2. Assessed by a multidisciplinary team as not a candidate for curative surgical resection.

  3. No absolute contraindications for the combined implantation of a biliary metallic stent and an ^125^I seeds strand (e.g., severe coagulation dysfunction, significant renal impairment, or uncontrolled serious cardiovascular/cerebrovascular diseases).

  4. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Obstructive jaundice attributable to benign etiology.
2. Presence of any absolute contraindication listed in the inclusion criteria.
3. Life expectancy estimated to be less than three months.
4. Unwillingness to participate in the study or provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Stent Patency Time | From the date of randomization/stent placement until the date of documented stent re-obstruction or death from any cause, whichever occurs first, assessed up to 24 months.
  The duration from the date of stent placement to the date of first documented stent re-obstruction (confirmed by imaging evidence of restenosis or occlusion). For patients who die without prior evidence of recurrent jaundice, the data will be censored at the date of death.
Overall Survival | From the date of randomization/stent placement until the date of death from any cause, assessed up to 24 months.
  The time from the date of the stent placement procedure until the date of death from any cause. For patients who are alive at the end of the study, survival data will be censored at the date of the last follow-up contact.

SECONDARY OUTCOMES:
Incidence of Procedure-Related Complications | Intraoperative period and up to 30 days after the procedure.
  The composite rate of intraoperative and postoperative adverse events. Assessed complications include nausea/vomiting, abdominal pain, hemobilia, vagus reflex, fever, biliary fistula, and biliary peritonitis. Each complication will be documented as present or absent based on clinical and diagnostic criteria.
Change in Serum Total Bilirubin (TBIL) Level | Baseline (pre-PTBSIS, after initial PTBD) and 1 month after the PTBSIS procedure.
  The absolute change in serum total bilirubin concentration (measured in μmol/L) from the pre-procedure baseline (after initial PTBD drainage) to 1 month after the combined stent and seed strand implantation procedure.
Change in Serum Alanine Aminotransferase (ALT) Level | Baseline (pre-PTBSIS, after initial PTBD) and 1 month after the PTBSIS procedure.
  The absolute change in serum alanine aminotransferase activity (measured in U/L) from the pre-procedure baseline (after initial PTBD drainage) to 1 month after the combined stent and seed strand implantation procedure.
Change in Serum Aspartate Aminotransferase (AST) Level | Baseline (pre-PTBSIS, after initial PTBD) and 1 month after the PTBSIS procedure.
  The absolute change in serum aspartate aminotransferase activity (measured in U/L) from the pre-procedure baseline (after initial PTBD drainage) to 1 month after the combined stent and seed strand implantation procedure.
Technical Success Rate | Assessed immediately upon completion of the stent and seed strand implantation procedure.
  The proportion of procedures in which both the biliary metallic stent and the ^125^I seeds strand are successfully and precisely deployed at the intended target lesion site, as confirmed by immediate post-procedure fluoroscopy demonstrating unobstructed flow of contrast medium through the stent lumen into the duodenum.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang W, Shen J, Wang C, Ren B, Zhu X, Ni C. Safety and Feasibility of Helical I-125 Seed Implants Combined with Transcatheter Arterial Chemoembolization in Hepatocellular Carcinomas with Main Portal Vein Tumor Thrombus. Cardiovasc Intervent Radiol. 2019 Oct;42(10):1420-1428. doi: 10.1007/s00270-019-02256-z. Epub 2019 Jun 11. PMID 31187228
- [Result] Jang S, Stevens T, Parsi MA, Bhatt A, Kichler A, Vargo JJ. Superiority of Self-Expandable Metallic Stents Over Plastic Stents in Treatment of Malignant Distal Biliary Strictures. Clin Gastroenterol Hepatol. 2022 Feb;20(2):e182-e195. doi: 10.1016/j.cgh.2020.12.020. Epub 2020 Dec 18. PMID 33346140
- [Result] Larghi A, Tringali A, Lecca PG, Giordano M, Costamagna G. Management of hilar biliary strictures. Am J Gastroenterol. 2008 Feb;103(2):458-73. doi: 10.1111/j.1572-0241.2007.01645.x. Epub 2007 Nov 19. PMID 18028506